CLINICAL TRIAL: NCT07162909
Title: The Time Before the Crime: Risk Patterns in Individuals Who Commit Criminal Acts and Undergo a Forensic Psychiatric Evaluation
Brief Title: The Time Before the Crime - Risk Patterns in Offenders Undergoing a Forensic Psychiatric Evaluation
Acronym: Tibec
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Katarina Howner, Associate professor, Karolinska Institutet
Other Study IDs: 2024-07566-01
Record Dates: First submitted 2025-06-23; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Crime
Keywords: severe mental disorder; forensic psychiatric evaluation; risk patterns; violence
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: The study population consists of individuals aged ≥ 18 years who have had or currently have contact with a psychiatric care provider within Region Stockholm (public clinic or private provider with a regional agreement) whose medical records were requested by the National Board of Forensic Medicine (NBFM) in 2023 for forensic psychiatric evaluation (§ 7-evaluation or FPE), estimated to be n=250.
- Controls: The control group consists of individuals aged ≥ 18 years who have had or currently have contact with a psychiatric care provider within Region Stockholm (public clinic or private provider with a regional agreement) whose medical records were not requested by the NBFM in 2023. The control group is matched to the study population based on gender, age and psychiatric care unit (psychiatric intensive care units, psychosis ward, general psychiatric ward, psychiatric outpatient clinic, psychiatric emergency unit). Thereby we hope that the control group will consist of individuals with similar psychiatric conditions and care burden as the study population.

SUMMARY:
The overarching aim of the research project is to identify risk patterns preceding criminal acts among individuals later subject to forensic psychiatric evaluation (FPE) in Sweden, including factors within psychiatric care as well as broader individual or contextual factors.

Although individuals who undergo an FPE represent a small subset of all individuals who commit criminal acts, the implications of being sentenced to forensic psychiatric care are profound. In Sweden, approximately 300 individuals are transferred to forensic psychiatric care each year, with a median duration of 7.5 years. Notably, the number of admissions exceeds the number of discharges annually, resulting in a growing forensic psychiatric population. This increasing trend underscores the need for increased knowledge and preventive efforts. All forensic psychiatric patients undergo an FPE before the sentencing, and previous studies show that most of these individuals were already known to the psychiatric system prior to the offenses, which means that individuals in these groups are overlapping. However, the mean length of stay in psychiatric inpatient compulsory care is much shorter than that in forensic psychiatric care. Clinical expertise from FPEs suggests that identifiable risk patterns may exist before the criminal offence. The question of whether such potential risk patterns exist within this patient group has not been systematically studied before, which is why the current study aims to investigate this issue. Can risk patterns be identified within psychiatric care prior to the offense? If risk patterns can be identified, knowledge of such risk patterns could hopefully increase risk awareness within psychiatric services and lead to more frequent and accurate violence risk assessments. Knowledge of such risk patterns could also serve as a foundation for preventive measures. The long-term goal is to reduce the likelihood that individuals receiving psychiatric care progress to becoming forensic psychiatric patients.

DETAILED DESCRIPTION:
Case-control study

Design and methodology:

The study is designed as a case-control study. The study population consists of individuals aged ≥ 18 years who have had or currently have contact with a psychiatric care provider within Region Stockholm (public clinic or private provider with a regional agreement) whose medical records were requested by the NBFM in 2023 for forensic psychiatric evaluation (§ 7-evaluation or FPE), estimated to be n=250.

The control group consists of individuals aged ≥ 18 years who have had or currently have contact with a psychiatric care provider within Region Stockholm (public clinic or private provider with a regional agreement) whose medical records were not requested by the NBFM in 2023. The control group is matched to the study population based on gender, age and psychiatric care unit (psychiatric intensive care units, psychosis ward, general psychiatric ward, psychiatric outpatient clinic, psychiatric emergency unit). Thereby we hope that the control group will consist of individuals with similar psychiatric conditions and care burden as the study population.

An exclusion criterion for the study population is if the offense underlying the NBFM request for the medical records (the index offense) occurred before 2018. This is because the study aims to investigate psychiatric care as it is currently structured and provided. An exclusion criterion for the control group is if the individual previously underwent an FPE at some point. Additional exclusion criteria for both groups are if there is no registered psychiatric care contact in Region Stockholm's shared electronic medical record system, TakeCare, three months prior to the date of the index offense.

The individuals whose medical records were requested by the NBFM in 2023 for forensic psychiatric evaluations (§ 7 evaluation or FPE) are identified by retrieving data from TakeCare. The NBFM's requests for medical records are documented routinely with a specific search term in TakeCare, minimizing the risk of missing data. Once the individuals in the study population are identified, their personal identification numbers (PINs) are sent to the NBFM. Based on the PINs, the NBFM retrieves the relevant dates of criminal offenses for each individua in the study population. Additional variables are also identified in the NBFM case management system, including criminal charges, prior convictions, information about substance use at the time of the offense, and court rulings. If an individual has committed multiple offenses, the most serious offense is selected, i.e., the one with the highest penal value. In cases of repeated offenses with similar penal value or multiple offenses within the same criminal charge category, the date of the first offense is chosen as the index crime.

The retrospective record review is conducted systematically based on a predefined review template containing 26 markers. Each marker has a specific definition. During the planning phase of the project, the project team received input from a reference group consisting of professionals from various areas within healthcare. The reference group participated in meetings during the project's planning phase. The development of the 26 markers in the review template was carried out in collaboration with the reference group to ensure that the markers are as relevant and specific as possible. The review period is set to three months prior to the date of the alleged offense, as this is considered the period in which there would be the greatest opportunity to design specific interventions. In the control group, the medical record review is based on the same month as the dates of the matched offenses.

ELIGIBILITY:
Inclusion criteria, case group:

* Age ≥ 18 years
* Contact with a psychiatric care provider within Region Stockholm
* Medical records requested by the NBFM in 2023 for forensic psychiatric evaluation

Inclusion criteria, control group:

* Age ≥ 18 years
* Contact with a psychiatric care provider within Region Stockholm
* Medical records NOT requested by the NBFM in 2023 for forensic psychiatric evaluation

Matching criteria:

* Gender (male/female)
* Age group (18-24, 24-39 and >39 years)
* Psychiatric care unit

Exclusion Criteria, general:

* No registered psychiatric care contact in Region Stockholm's shared electronic medical record system, three months prior to the date of the index offense.

Exclusion Criteria, case group:

* The index offense before 2018.

Exclusion Criteria, control group:

* Individual previously underwent an FPE at some point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case group: individuals ≥ 18 years who had contact with at least one psychiatric care provider within Region Stockholm, Sweden. This included both clinics operated by a Swedish healthcare region and private clinics operating under regional agreements. Individuals eligible for the case group were those whose psychiatric medical records were requested by the Swedish National Board of Forensic Medicine (NBFM) in 2023 for the purpose of conducting a forensic psychiatric evaluation, either a preliminary assessment (§7 examination) or a full forensic psychiatric evaluation (FPE).
  Control group: Similar individuals, but whose psychiatric medical records were not requested by the NBFM in 2023 for the purpose of conducting a forensic psychiatric evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk markers | All risk makers will be searched for in the three-month period before the date of the criminal act (case croup) and also in a three-month period for the control group.
  26 predefined risk markers that will be searched for in the retrospective record review. All risk markers have their own specific definition. For detailed description, see attached document.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol: Review Template for TiBeC Medical Record Review (2025-08-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT07162909/Prot_000.pdf
  • Study Protocol: Variables for Review of Section 7 and FPEs (2025-08-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT07162909/Prot_001.pdf
  • Statistical Analysis Plan (2025-08-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT07162909/SAP_002.pdf